CLINICAL TRIAL: NCT02213393
Title: Effectiveness of Cater With Care Products in Reaching Recommendations for Protein Intake During and After Hospital Stay and in Improving Functional Status After Hospital Stay in Elderly Patients.
Brief Title: Cater With Care Effect Study
Acronym: CwC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL48893.081.14
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Undernutrition
Keywords: undernutrition; nutritional status; elderly patients; protein; enriched products; recovery; physical function; quality of life; activities of daily living
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protein enriched products (Experimental): The intervention group receives protein enriched products (CwC products) in the hospital and receives these also after discharge during 12 weeks.
  Interventions: Dietary Supplement: Protein enriched products
- Usual menu (Active Comparator): The control group receives the usual protein and energy rich menu in the hospital and receives regular products, no protein enrichment, after discharge during 12 weeks.
  Interventions: Dietary Supplement: Usual menu

INTERVENTIONS:
Dietary Supplement: Protein enriched products — The intervention group receives CwC protein enriched products. After discharge the intervention group receives CwC products delivered at home for 12 weeks.
  Other Names: CwC products
  Arms: Protein enriched products
Dietary Supplement: Usual menu — The control group receives the usual menu, which is energy and protein rich in this elderly patient group. After discharge the control group receives regular products, no protein enrichment, at home for 12 weeks.
  Arms: Usual menu

SUMMARY:
The objective is to study the effectiveness of supplementing a standard hospital and 12-week home menu with protein-enriched Cater with Care products in reaching a protein intake of 1,2-1,5 g/kg body weight/day and in improving functional status after hospital stay in elderly patients.

DETAILED DESCRIPTION:
Rationale: About 25% of hospitalized elderly patients are at risk of undernutrition at admission. Many hospitals provide an energy and protein enriched diet, extra snacks, and oral nutritional supplements if needed. Still, a considerable part of these patients are unable to meet protein requirements and are still at risk of undernutrition at hospital discharge. This may impair recovery of illness, partly due to loss of muscle mass and physical performance. To improve protein intake, Cater with Care products have been developed: a selection of foods and drinks that are consumed often by elderly persons, but now enriched with protein up to 10 grams per portion. We hypothesize that these products help to reach protein requirements in elderly patients during and after hospital stay and thereby improve their health outcomes.

Objective: To study the effectiveness of supplementing a standard hospital and 12-week home menu with protein-enriched Cater with Care products in reaching a protein intake of 1,2-1,5 g/kg/day and in improving functional status after hospital stay in elderly patients.

Study design: Randomised Controlled Trial (RCT) with 2 intervention groups and two phases: a hospital phase including all admitted patients and a home phase with a selection of patients.

Study population: Patients of 65 years or over who are admitted to the departments of Geriatrics, Pulmonary Disease, or Internal Medicine of Hospital Gelderse Vallei.

Intervention: The control group receives the standard hospital menu for elderly at risk of undernutrition (energy and protein rich) and a variety of foods and drinks to be used as part of their home diet for 12 weeks after hospitalization. Foods and drinks for home use are non-enriched variants of Cater with Care products (e.g. normal fruit juice).

The intervention group receives Cater with Care protein-enriched foods and drinks during hospital stay (in addition to the standard hospital menu) and at home as part of their home diet for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hospital phase:
* admitted to the wards of Geriatric medicine, Pulmonary Medicine, or Internal Medicine in Hospital Gelderse Vallei
* aged 65 years or over
* being eligible for receiving a standard protein enriched menu based on hospital protocol
* Home phase:
* included in the hospital phase of the study
* consent to continue treatment and study participation after hospital discharge

Exclusion Criteria:

* Hospital phase:
* unwilling to give consent for gathering data from the medical record or meal service system
* unable to understand Dutch
* food allergies, food intolerances or other dietary restrictions that prevents the patient from receiving the standard protein enriched menu or Cater with Care products based on the judgement of a dietician and/or medical staff
* expected length of hospital stay less than 4 days
* renal insufficiency (eGFR < 30 ml/min)
* starting with tube feeding or total parenteral nutrition within 2 days of admission
* refeeding syndrome score > 0 based on hospital screening tool for refeeding risk
* delirium at admission
* receiving palliative care
* Home phase:
* going to a nursing home, rehabilitation centre or hospice after hospital discharge
* cognitive impairment or diagnosed with dementia
* legally incapacitated

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Protein intake and Physical functioning at 6 months | 6 months
  This study has 2 primary outcomes: protein intake and physical functioning. These will be assessed at baseline (0), and 2, 6, 12 and 24 weeks after hospital discharge.

SECONDARY OUTCOMES:
Change in muscle strength from baseline to 6 months. | 6 months
  Muscle strength (leg and hand grip) will be assessed at baseline (0), and 2, 6, 12 and 24 weeks after hospital discharge.
Change in nutritional status from baseline to 6 months. | 6 months
  Nutritional status (MNA and dietary intake) will be assessed at baseline (0), and 2, 6, 12 and 24 weeks after hospital discharge.
Change in Quality of Life from baseline to 6 months. | 6 months.
  Quality of Life will be assessed with the EuroQoL-5D-5L (at baseline, and 12 and 24 weeks after hospital discharge)
Change in Activities of Daily Living from baseline to 6 months. | 6 months
  Activities of Daily Living (ADL) will be assessed by using the Barthel index (at baseline, and 2, 6, 12 and 24 weeks after hospital discharge).

OTHER OUTCOMES:
BMI | 6 months
  BMI is calculated from weight and length measurements at baseline (0), 2, 6, 12, 24 weeks after hospital discharge.
Physical Activity | 6 months
  Physical Activity will be assessed by using the LAPAQ questionnaire.
Length of hospital stay | 12 weeks
  The length of hospital stay will be recorded to include in an economic evaluation.
Costs of hospital stay | 12 weeks
  After discharge from the hospital, the costs of hospital stay will be calculated to include in the economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M de Roos, PhD, Principal Investigator — Wageningen University
Locations (1):
- Hospital Gelderse Vallei, Ede, Gelderland, Netherlands

REFERENCES:
- [Derived] Beelen J, Vasse E, Janssen N, Janse A, de Roos NM, de Groot LCPGM. Protein-enriched familiar foods and drinks improve protein intake of hospitalized older patients: A randomized controlled trial. Clin Nutr. 2018 Aug;37(4):1186-1192. doi: 10.1016/j.clnu.2017.05.010. Epub 2017 May 18. PMID 28571713